CLINICAL TRIAL: NCT06910709
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose and Food-effect Study to Evaluate the Safety, Tolerability, Pharmacokinetics of AMG 378 in Healthy Participants
Brief Title: Single and Multiple Ascending Dose Study of AMG 378 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 20230274
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: The food-effect cohort will have a cross-over design with 2 periods.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Single Ascending Dose (SAD) (Experimental): Participants will be randomized in a 3:1 ratio to receive a single dose of either AMG 378 or placebo.
  Interventions: Drug: AMG 378; Drug: Placebo
- Part A: Food-effect Cohort (Experimental): Participants will be randomized 1:1 in a cross-over design to receive a single dose of AMG 378 in each of the 2 periods. Dosing under fasting conditions will occur after a 10-hour fast. Dosing under fed conditions will be within 30 minutes of the start of a high-fat breakfast. There will be a 7-day washout between each cross-over period.
  Interventions: Drug: AMG 378
- Part B: Multiple Ascending Dose (MAD) (Experimental): Participants will be randomized in a 3:1 ratio to receive multiple doses of either AMG 378 or placebo.
  Interventions: Drug: AMG 378; Drug: Placebo

INTERVENTIONS:
Drug: AMG 378 — Oral tablet
Drug: Placebo — Oral tablet
  Arms: Part A: Single Ascending Dose (SAD); Part B: Multiple Ascending Dose (MAD)

SUMMARY:
The main objective of the study is to assess the safety and tolerability of AMG 378 as single or multiple doses in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 to ≤ 55 years (inclusive) at the time of signing the informed consent.
* Body mass index between 18 and 30 kg/m^2, inclusive, at screening.
* Men (even with a history of vasectomy) with partners of childbearing potential must agree to practice sexual abstinence or use a male barrier method of contraception (ie, male condom with spermicide) in addition to a second method of acceptable contraception by female partner from Check-in until 30 days after the last dose of investigational product.
* Participant must be overtly healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, vital signs, physical examination, laboratory tests, and 12-lead electrocardiogram (ECG) recording(s) at the screening and Day 1 visits.

Exclusion Criteria:

* History of malignancy of any type.
* History of esophageal, gastric, or duodenal ulceration prior to screening visit.
* Evidence of active bacterial, viral, fungal or parasitic infections within the last 30 days prior to study Day 1.
* History or evidence of clinically significant arrhythmia at screening, or Day 1 ECG.
* A QT interval corrected for heart rate (HR) based on the Fridericia method (QTcF) interval > 450 ms in all participants regardless of biological sex or history/evidence of long QT syndrome at screening or study Day -1.
* Positive results for human immunodeficiency virus (HIV) antibodies, HIV antigen, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C virus ribonucleic acid (RNA) at screening.
* History of active tuberculosis (TB) infection, current symptoms concerning for active TB, or positive or indeterminate interferon gamma release assay (IGRA).
* Positive test for drugs, cotinine (tobacco use) or alcohol use at screening or on Day -1.
* Sexually active female participants of childbearing potential unwilling to use 2 protocol specified highly effective methods of contraception during treatment and for an additional 30 days after the last dose of investigational product.
* Alcohol consumption from 48 hours prior to study Day 1.
* Use of tobacco- or nicotine-containing products within 6 months prior to study Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing a Treatment-emergent Adverse Event (TEAE) | Day 1 to Day 30 (SAD/MAD) or Day 40 (food effect cohort)

SECONDARY OUTCOMES:
SAD/MAD Only: Maximum Observed Concentration (Cmax) of AMG 378 | Day 1 to Day 30
SAD/MAD Only: Time of Cmax (Tmax) of AMG 378 | Day 1 to Day 30
SAD/MAD Only: Area Under the Concentration Time Curve (AUC) of AMG 378 | Day 1 to Day 30
Food Effect Cohort Only: AUC of AMG 378 in the Fed Versus Fasted State | Day 1 to Day 14
Food Effect Cohort Only: Cmax of AMG 378 in the Fed Versus Fasted State | Day 1 to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Orange County Research Center, Lake Forest, California
  - Dr. Vince Clinical Research, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com